CLINICAL TRIAL: NCT03124342
Title: Vanderbilt ICU Recovery Program Pilot Trial
Acronym: VIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Matthew Semler, Assistant Professor of Medicine, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 170126
Record Dates: First submitted 2017-04-18; First posted 2017-04-21 (Actual); Results first posted 2019-10-08 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Intensive Care Unit Syndrome; Intensive Care Neurological Disorder; Intensive Care (ICU) Myopathy; Intensive Care Psychiatric Disorder (Diagnosis)
MeSH Terms: conditions — Muscular Diseases; Disease | interventions — Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VANDERBILT ICU RECOVERY PROGRAM (VIP) (Experimental): Patients assigned to the Vanderbilt ICU Recovery Program (VIP) group will receive the components of the ICU Recovery Program intervention.
  Interventions: Other: VANDERBILT ICU RECOVERY PROGRAM
- Usual care (No Intervention): Patients in the usual care group will receive care as dictated by their clinical team. In usual care in the study institution, patients frequently receive medication reconciliation by and ICU pharmacist at the time of transfer out of the ICU to the hospital ward, medication reconciliation by a physician at the time of hospital discharge, and follow up with their primary care physician within two weeks of hospital discharge. Usual care does not currently include an in-person assessment of the patient's cognitive and functional status or anticipated post-ICU needs by a nurse practitioner between ICU transfer and hospital discharge, access to a 24/7 contact line after hospital discharge, or assessment in a multi-disciplinary ICU Recovery Clinic.

INTERVENTIONS:
Other: VANDERBILT ICU RECOVERY PROGRAM — 10-component ICU Recovery Program intervention, including:
  1. Nurse Practitioner In-Person Visit at the time of transfer from the ICU
  2. Provision of an ICU Recovery Program Pamphlet describing post-intensive care syndrome and providing online resources
  3. Performance of formal medication reconciliation at the time of transfer from the ICU
  4. Access to a dedicated 24-hour a day, 7-day a week contact line
  5. ICU Recovery Clinic Visit Medical Examination.
  6. ICU Recovery Clinic Medication Reconciliation and Counseling
  7. ICU Recovery Clinic Cognitive/Mental Health Assessment and Psychoeducation. A brief session of psychotherapy conducted by a clinical psychologist
  8. ICU Recovery Clinic Case Management. A brief case management consultation
  9. ICU Recovery Clinic Patient Centered Consultation. A final consultation with patients and families by a PCCM physician
  10. Directed Subspecialty Referrals
  Other Names: Intervention
  Arms: VANDERBILT ICU RECOVERY PROGRAM (VIP)

SUMMARY:
Every year, millions of Americans are admitted to the intensive care unit. Due to advances in critical care, mortality rates are decreasing, increasing the number of ICU survivors. Survivors of critical illness, however, often face physical, functional, and cognitive deficits that place them at risk for a cycle of re-hospitalization that frequently culminates in premature death. Moreover, post-ICU interventions may be resource-intensive and may be most cost-effective only in a subgroup of patients at highest risk. Whether a multi-disciplinary program to facilitate recovery from critical illness can prevent hospital readmission and improve quality of life among high-risk ICU survivors remains unknown. The primary aim of this pilot is to examine the feasibility of implementing a multidisciplinary ICU Recovery Program and the influence of such a program on process measures including contact with the ICU recovery team and attendance of ICU recovery clinic. The secondary aims are to compare the effect of an ICU Recovery Program on 30-day same-hospital readmission and other clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Admitted to the Medical Intensive Care Unit (MICU) at Vanderbilt University Medical Center for at least 48 hours
3. Estimated risk of 30-day same-hospital readmission greater than 15%
4. Not previously enrolled in the study.

Exclusion Criteria:

1. Long-term residence at a skilled nursing facility
2. Long-term mechanical ventilation prior to admission
3. Solid organ or stem cell transplantation
4. Recorded primary residency > 200 miles from Vanderbilt
5. Comfort care only

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2018-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Stollings, PharmD, Study Director — Vanderbilt University Medical Center; Carla Sevin, MD, Study Chair — Vanderbilt University Medical Center; Matthew W Semler, MD, MSc, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- VANDERBILT ICU RECOVERY PROGRAM (VIP): VANDERBILT ICU RECOVERY PROGRAM -- 10-component ICU Recovery Program intervention, including:
  1. Nurse Practitioner In-Person Visit at the time of transfer from the ICU
  2. Provision of an ICU Recovery Program Pamphlet describing post-intensive care syndrome and providing online resources
  3. Performance of formal medication reconciliation at the time of transfer from the ICU
  4. Access to a dedicated 24-hour a day, 7-day a week contact line
  5. ICU Recovery Clinic Visit Medical Examination.
  6. ICU Recovery Clinic Medication Reconciliation and Counseling
  7. ICU Recovery Clinic Cognitive/Mental Health Assessment and Psychoeducation. A brief session of psychotherapy conducted by a clinical psychologist
  8. ICU Recovery Clinic Case Management. A brief case management consultation
  9. ICU Recovery Clinic Patient Centered Consultation. A final consultation with patients and families by a PCCM physician
  10. Directed Subspecialty Referrals
Period: Overall Study
Arm/Group | VANDERBILT ICU RECOVERY PROGRAM (VIP) | Usual Care
Started | 111 | 121
Completed | 111 | 121
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VANDERBILT ICU RECOVERY PROGRAM (VIP) | Usual Care | Total
Number analyzed (Participants) | 111 | 121 | 232
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 56 [44 to 67] | 56 [48 to 66] | 56 [46 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 54 | 114
  Male | 51 | 67 | 118
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 21 | 20 | 41
  White | 83 | 89 | 172
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 12 | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Components of the ICU Recovery Program Received
Description: Number of components of the ICU Recovery Program intervention received by patients between ICU transfer and 30 days after hospital discharge. The 10-components considered part of the ICU Recovery Program include: (1) nurse practitioner in-person visit between ICU transfer and hospital discharge, (2) ICU Recovery Program pamphlet, (3) pharmacist medication reconciliation at the time of ICU transfer, (4) ICU Recovery Program contact line, (5) nurse practitioner history and physical in ICU Recovery Clinic, (6) pharmacist medication reconciliation in ICU Recovery Clinic, (7) cognitive/mental health assessment and psychoeducation in ICU Recovery Clinic, (8) case management consultation in ICU Recovery Clinic, (9) patient centered consultation with pulmonary and critical care medicine physician in ICU Recovery clinic, (10), directed subspecialty referrals.
Time Frame: From the time of study enrollment to 30 days after hospital discharge
Measure: Median (Inter-Quartile Range); unit: interventions
Arm/Group | VANDERBILT ICU RECOVERY PROGRAM (VIP) | Usual Care
Number analyzed (Participants) | 111 | 121
interventions | 2 [1 to 3] | 1 [0 to 1]

2. Secondary Outcome: Number of Participants With Same-hospital Readmission in the 30 Days After Hospital Discharge
Description: Readmission to the study hospital in the 30 days after hospital discharge
Time Frame: Within 30 days of hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | VANDERBILT ICU RECOVERY PROGRAM (VIP) | Usual Care
Number analyzed (Participants) | 111 | 121
Participants | 16 | 26

3. Secondary Outcome: Number of Participants Death or Readmission in the 30 Days After Hospital Discharge
Description: Composite outcome of death or readmission in the 30 days after hospital discharge
Time Frame: Within 30 days of hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | VANDERBILT ICU RECOVERY PROGRAM (VIP) | Usual Care
Number analyzed (Participants) | 111 | 121
Participants | 20 | 36

4. Secondary Outcome: Number Participants With Same-hospital Emergency Department Visits in the 30 Days After Hospital Discharge
Time Frame: Within 30 days of hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | VANDERBILT ICU RECOVERY PROGRAM (VIP) | Usual Care
Number analyzed (Participants) | 111 | 121
Participants | 1 | 1

5. Secondary Outcome: Number of Same-hospital Outpatient Clinic Visits in the 30 Days After Hospital Discharge
Time Frame: Within 30 days of hospital discharge
Measure: Number; unit: visits
Groups:
- VANDERBILT ICU RECOVERY PROGRAM (VIP): Patients assigned to the Vanderbilt ICU Recovery Program (VIP) group will receive the components of the ICU Recovery Program intervention.
  VANDERBILT ICU RECOVERY PROGRAM: 10-component ICU Recovery Program intervention, including:
  1. Nurse Practitioner In-Person Visit at the time of transfer from the ICU
  2. Provision of an ICU Recovery Program Pamphlet describing post-intensive care syndrome and providing online resources
  3. Performance of formal medication reconciliation at the time of transfer from the ICU
  4. Access to a dedicated 24-hour a day, 7-day a week contact line
  5. ICU Recovery Clinic Visit Medical Examination.
  6. ICU Recovery Clinic Medication Reconciliation and Counseling
  7. ICU Recovery Clinic Cognitive/Mental Health Assessment and Psychoeducation. A brief session of psychotherapy conducted by a clinical psychologist
  8. ICU Recovery Clinic Case Management. A brief case management consultation
  9. ICU Recovery Clinic Patient Centered Consultation.
Arm/Group | VANDERBILT ICU RECOVERY PROGRAM (VIP) | Usual Care
Number analyzed (Participants) | 111 | 121
visits | 14 | 0

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | VANDERBILT ICU RECOVERY PROGRAM (VIP) | Usual Care
All-Cause Mortality (participants affected / at risk) | 7/111 | 10/121
Serious Adverse Events (participants affected / at risk) | 0/111 | 0/121
Other Adverse Events (participants affected / at risk) | 0/111 | 0/121

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-12): https://cdn.clinicaltrials.gov/large-docs/42/NCT03124342/Prot_SAP_000.pdf